CLINICAL TRIAL: NCT00559247
Title: Placebo-Controlled Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of BMS-650032 in Subjects Chronically Infected With Hepatitis C Virus Genotype 1
Brief Title: A Single Ascending Dose Study of BMS-650032 in HCV Infected Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AI447-002
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — asunaprevir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- or Placebo - Dose Panel 1 (Experimental): Oral Suspension, 10 mg
  Interventions: Drug: BMS-650032 or Placebo
- or Placebo - Dose Panel 2 (Experimental): Oral Suspension 50 mg
  Interventions: Drug: BMS-650032 or Placebo
- or Placebo - Dose Panel 3 (Experimental): Oral Suspension, 200 mg
  Interventions: Drug: BMS-650032 or Placebo
- or Placebo - Dose Panel 4 (Experimental): Oral Suspension or Solution, 2.5 to 600 mg
  Interventions: Drug: BMS-650032 or Placebo

INTERVENTIONS:
Drug: BMS-650032 or Placebo — Oral, Once daily, Single Dose

SUMMARY:
The primary purpose of this study is to evaluate the safety profile and tolerability of single oral doses of BMS-650032 in subjects with chronic hepatitis C infection

ELIGIBILITY:
Inclusion Criteria:

* Chronically infected with HCV genotype 1
* Treatment naive or treatment non-responders or treatment intolerant
* HCV RNA viral load of ≥10*5 IU/mL
* BMI 18 to 35kg/m²

Exclusion Criteria:

* Any significant acute or chronic medical illness which is not stable or is not controlled with medication and not consistent with HCV infection
* Major surgery within 4 weeks of study drug administration and any gastrointestinal surgery that could impact the absorption of study drug
* Co-infection with HIV or HBV
* Women of childbearing potential

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Safety Outcome Measures | Safety and tolerability assessments will be performed for a period of 7 days after administration of a single dose

SECONDARY OUTCOMES:
Pharmacokinetic Measures | Pharmacokinetic assessments will be done for a period of 72 hours following administration of a single oral dose
Pharmacodynamic Measures | Antiviral activity will be assessed by the magnitude and rate of change in plasma HCV RNA levels for a period of 7 days after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (5):
  - West Coast Clinical Trials, Llc, Cypress, California
  - Orlando Clinical Research Center, Orlando, Florida
  - Parexel International Corporation, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Alamo Medical Research, San Antonio, Texas